CLINICAL TRIAL: NCT04716478
Title: Creation of a Prospective Endodontics Database
Brief Title: Prospective Endodontics Database
Acronym: REone
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL20_0833
Record Dates: First submitted 2021-01-15; First posted 2021-01-20 (Actual); Last update posted 2021-05-06 (Actual); Status verified 2021-01

CONDITIONS: Apical Periodontitis
MeSH Terms: conditions — Periapical Periodontitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient in need of endodontic care
  Interventions: Other: Clinical and radiological data collection

INTERVENTIONS:
Other: Clinical and radiological data collection — No specific intervention. Data of the usual care will be collected as the demographic data, the medical history, imaging report, etc.

SUMMARY:
Endodontic treatment is necessary after certain dental trauma or in the presence of a large carious lesion, associated with signs of irreversible pulpal inflammation. The treatment of apical periodontitis is a real public health issue. The endodontic success rate is between 68 and 85%. Indeed, some studies show that systemic diseases such as diabetes can increase the prevalence and bone loss associated with apical periodontitis. Other studies identify apical periodontitis as a factor that can potentiate symptoms caused by inflammatory diseases such as cardiovascular disease and diabetes by increasing the level of inflammatory cells in the blood.

However, since 2014 the European Society of Endodontology has recommended establishing a higher level of evidence to ensure the link that these pathologies may have. For this, it is necessary to assess the criteria that may influence the healing of apical periodontitis.

Endodata has been developed by dental surgeons specializing in endodontics. The purpose of this software is to improve the clinical follow-up of patients and to establish a clinical and radiological database. In this context, the creation of a clinical database including data for all root canal treatment is of high interest.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient aged ≥ 18,
* New patients received in consultation by students registered for a Diploma in Endodontics in one of the participating centres (Brest, Bordeaux, Lyon, Nancy, Nantes, Nice, Paris, Toulouse) or received by one of the private practitioners participating in the study;
* Patient with an indication for endodontic treatment or endodontic retreatment on at least one permanent tooth.

Exclusion Criteria:

* Patient unable to understand the purpose and conduct of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patient with apical periodontitis
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2021-01-22 (Actual); Primary Completion 2022-06-01 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
The main objective is to build a database with the necessary, relevant and quality data that will allow the development of a diagnostic and therapeutic aid in endodontics. | follow-up at 6 months.
  The patient's medical pathologies, the results of tests and clinical examination, radiological analysis and diagnostics is recorded during routine care. The treatment protocol is detailed for each technique, product or material used.

CONTACTS AND LOCATIONS:
Locations (21):
- France (21):
  - CHU de Bordeaux, Service de Médecine Buccodentaire, Bordeaux
  - CHU de Brest, Service d'Odontologie, Brest
  - Cabinet du Dr Baptiste Rivory, Lyon
  - Cabinet du Dr Matthieu Durand, Lyon
  - Cabinet du Dr Oussama Bouamar, Lyon
  - Cabinet du Dr Paul-Marie Oliva, Lyon
  - Hospices Civils de Lyon, Service d'Odontologie, Lyon
  - UFR d'Odontologie, Laboratoire des Multimatériaux et Interfaces, Lyon
  - CHRU de Nancy, Service d'Odontologie, Nancy
  - CHU de Nantes, Service d'Odontologie, Nantes
  - Cabinet du Dr Catherine Ricci, Nice
  - Assistance Publique des Hôpitaux de Paris, Hôpital Bretonneau, Service d'Odontologie, Paris
  - Assistance Publique des Hôpitaux de Paris, Hôpital Charles Foix, Service d'Odontologie, Paris
  - Assistance Publique des Hôpitaux de Paris, Hôpital Henri Mondor, Service d'Odontologie, Paris
  - Assistance Publique des Hôpitaux de Paris, Hôpital Pitié Salpêtrière, Service d'Odontologie, Paris
  - Cabinet du Dr Cauris Couvrechel, Paris
  - Cabinet du Dr Francois Bronnec, Paris
  - Cabinet du Dr Sandrine Dahan, Paris
  - Cabinet du Dr Valentin Marchi,, Paris
  - CHU de Toulouse, Service d'Odontologie, Toulouse
  - Cabinet du Dr Stéphanie Lapon, Tours